CLINICAL TRIAL: NCT01908517
Title: A Randomized Longitudinal Intervention Study to Assess Whether Electronic Messaging Can Increase Human Papilloma Viruses (HPV) Vaccine Utilization and Adherence Among Adolescents in Eastern North Carolina.
Brief Title: Human Papilloma Viruses (HPV) Vaccine Adherence Community Clinic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Essie Torres, Assistant Professor, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Merck-50915
Record Dates: First submitted 2013-07-15; First posted 2013-07-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Patient Compliance
Keywords: HPV Vaccine Adherence; Electronic Reminders
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPV Vaccine Electronic Reminders (Experimental): Parents in the intervention group will receive 1 electronic message per month in addition to the baseline and final assessments which equates to 8 contacts over a 7 month period. Specifically, intervention group participants will receive 4 education messages, 2 reminder/education messages, as well as 1 baseline and 1 final assessment survey.
  Interventions: Behavioral: HPV Vaccine Electronic Reminders

INTERVENTIONS:
Behavioral: HPV Vaccine Electronic Reminders — The intervention group will receive 4 education messages, 2 reminder/education messages, as well as 1 baseline and 1 final assessment survey. Control group participants will receive 2 contacts throughout the study, 1 at baseline and 1 at their final assessment survey. Up to two reminder contacts will be used if surveys are not completed for both intervention and control group participants. Preference for receipt of reminders will be obtained from the information study card parents complete at study enrollment. Enrollment card content, educational messages and patient- reminders will all be developed with community input.

SUMMARY:
There has been very limited research that has looked at electronic reminders (text messages) and its effectiveness in adherence to vaccination among low-income minority populations. Results have shown that text messages, among low-income parents and adolescents who were identified as having a cellphone, is an effective strategy to increase the likelihood of adolescent vaccination adherence. Hard copy and electronic messaging reminders have also been proven to be effective when coupled with other prevention strategies for immunizations for influenza and pneumococcal pneumonia and screening for colon, breast, and cervical cancer in adults. Additionally, Merck and Co. recommend electronic reminders in their patient compliance program as a key strategy for adherence. To our knowledge, this community-based pilot intervention study will be the first to assess electronic reminders and HPV vaccine initiation and adherence among rural uninsured and Medicaid populations. The investigators hypothesize that adolescent whose parents who receive the intervention will be more likely to initiate HPV vaccination and be compliant at 3 months and at 7 months as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Caretaker has Medicaid or is Uninsured
* Parent/Caretaker has a child between 11- 18 y/o
* Parent/Caretaker should be able to read English or Spanish
* Parent/Caretaker should have a phone and/or email address to provide for the study

Exclusion Criteria:

* Parents who have children younger than 11 or older than 18 years of age
* Parents who are not currently uninsured or enrolled in Medicaid/Medicare.
* Parent/Caretaker's child who received the 1st dose of HPV vaccine before enrolling in study

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 522 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Vaccine Adherence, as measure by receiving the 3 recommended doses withing a 6 month time period. | 7 months after initial HPV Vaccince shot
  Vaccine adherence will be measured using the CDC's guidelines which state that the second dose be given one to two months after the first, and the third dose be given six months after the first dose.

SECONDARY OUTCOMES:
HPV Knowledge, as measured by a 20% increase in knowledge about HPV and HPV vaccine among the intervention group. | 7 months after the first initial HPV vaccine shot
  Parents in the intervention group will receive 4 tailored education messages and 2 tailored reminder/education messages within the 6 month window period for the recommended HPV vaccine adherence guidelines. In order to assess a 20% increase in knowledge about HPV and the HPV vaccine, parents will take a baseline assessment survey and then a final assessment survey at the 7-month point once the vaccine series is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Essie Torres, PhD, MPH, Principal Investigator — East Carolina University; Alice Richman, PhD, MPH, Principal Investigator — East Carolina University
Locations (2):
- United States (2):
  - East Carolina University's General Pediatric Outpatient Clinic, Greenville, North Carolina
  - Kate B. Reynolds Medical Center, Snow Hill, North Carolina

REFERENCES:
- [Derived] Richman AR, Torres E, Wu Q, Carlston L, O'Rorke S, Moreno C, Olsson J. Text and Email Messaging for Increasing Human Papillomavirus Vaccine Completion among Uninsured or Medicaid-insured Adolescents in Rural Eastern North Carolina. J Health Care Poor Underserved. 2019;30(4):1499-1517. doi: 10.1353/hpu.2019.0090. PMID 31680111